CLINICAL TRIAL: NCT03930875
Title: Aspirin Resistance in Obstructive Sleep Apnea Patients (ARISA Trial)
Brief Title: Aspirin Resistance in OSA Patients
Status: Completed | Type: Observational
Sponsor: Danbury Hospital (Other)
Collaborators: Accriva Diagnostics (Industry)
Responsible Party: Principal Investigator, Jose Luis Mendez, Physician, Department of Pulmonary, Danbury Hospital
Other Study IDs: 17-08-229-337
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control - No Obstructive Sleep Apnea with Aspirin: The control group consist of patients with a negative diagnosis of OSA (based on a negative home sleep apnea test (REI) < 5 and attended sleep study, AHI < 5; or attended NPSG with an AHI < 5) and the patient is taking aspirin at a dose of 81 mg/day for at least a week prior to inclusion.
  After obtaining written informed consent, approximately 6 ml of blood was collected via venipuncture.
  Interventions: Other: Aspirin Resistance testing
- Arm 1- Obstructive Sleep Apnea with CPAP therapy and Aspirin: Arm 1 consist of patients with a diagnosis of OSA (based on home or attended sleep study) with an REI/AHI > 15 with or without symptoms or REI/AHI > 5 with symptoms of sleep apnea in a patient 18-85 years old, CPAP has been started within the last 2 years, and patient is taking aspirin at a dose of 81mg/day for at least a week, last dose taken within 24 hours prior to enrollment.
  After obtaining written informed consent, approximately 6 ml of blood was collected via venipuncture.
  Interventions: Other: Aspirin Resistance testing
- Arm 2 -Obstructive Sleep Apnea with no CPAP & Aspirin: Arm 2 consist of patients with a diagnosis of OSA (based on home or attended sleep study) with an REI/AHI > 15 with or without symptoms or REI/AHI > 5 with symptoms of sleep apnea in a patient 18-85 years old and patient is taking aspirin at a dose of 81mg/day for at least a week, last dose taken within 24 hours prior to enrollment.
  After obtaining written informed consent, approximately 6 ml of blood was collected via venipuncture.
  Interventions: Other: Aspirin Resistance testing

INTERVENTIONS:
Other: Aspirin Resistance testing — Aspirin resistance will be measured using platelet aggregometry (VerifyNow assay)

SUMMARY:
Obstructive Sleep Apnea (OSA) patients are at increased risk of major cardiovascular events, so many patients take aspirin for prevention. Poor responsiveness to aspirin is a major clinical concern because it can potentially worsen the prognosis of OSA patients. However, continuous positive airway pressure (CPAP) therapy that is considered standard of care for OSA treatment may potentially lead to improvement in responsiveness to aspirin. This study will determine whether CPAP therapy decreases patients' aspirin resistance in OSA patients with a new diagnosis or existing moderate to severe OSA who are treated with CPAP and take aspirin for prevention.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is a common sleep-related breathing disorder that afflicts more than 25 million adults in the United States. This number continues to rise yearly due to increased incidence of obesity in the United States. The prevalence of OSA among males and females is also on the rise with 34% of males and 17% of females diagnosed with this disease.

OSA is characterized as intermittent pharyngeal soft-tissue obstruction due to anatomical or positional etiology during sleep. This leads to episodes of hypoxemia and apneas which result in overall sleep fragmentation. The pathophysiology associated with OSA is complex. However, some proposed causes of OSA include hypoxia during sleep which causes increased circulating catecholamines and sympathetic activation, free radical formation leading to oxidative stress, increased cytokine release and endothelial dysfunction. These proposed mechanisms are also associated with increased platelet aggregation and hyperactivity and increase a patient's overall risk for cardiovascular morbidities.

Many patients with cardiovascular co-morbidities are taking aspirin for primary or secondary prevention. With a concomitant diagnosis of OSA, it is thought that these patients who are taking aspirin on a daily basis may become resistant to its effects based on how their OSA is controlled (ie. CPAP vs. Non-CPAP). Although aspirin resistance has been noted to be a "laboratory phenomenon," there have been studies which have shown a three-fold increase in cardiovascularco- morbidities in patients who were found to be aspirin resistant. In this study, it is our goal to determine the prevalence of aspirin resistance in patients who have a diagnosis of OSA and undergoing treatment with CPAP or Non-CPAP methods by measuring Aspirin Resistant Units (ARUs) using light aggregometry. It is our overall objective to determine whether or not OSA is an independent risk factor for aspirin resistance.

OSA patients are at increased risk of major cardiovascular events and aspirin resistance is associated with poor cardiovascular outcomes. Studying aspirin responsiveness in OSA patients may help to elucidate the potential role of platelet function testing, including the possible clinical implications of an aspirin therapy regimen guided by platelet function testing.

ELIGIBILITY:
Inclusion Criteria for Control Group:

* No OSA (based on home or attended polysomnography) determined by negative sleep study (HSAT or NPSG) REI/AHI < 5 (if a home study was done and found negative or equivocal an attended study is required to rule out sleep apnea)
* Patient is taking aspirin at a dose of 81 mg/day for at least a week last dose taken within 24 hours prior to enrollment.

Inclusion Criteria for "CPAP-Naïve" Cohort:

* Diagnosis of OSA (based on home or attended sleep study) with an REI/AHI ≥ 15 with or without symptoms or REI/AHI ≥ 5 with symptoms of sleep apnea in a patient 18-85 years old.
* Patient is taking aspirin at a dose of 81mg/day for at least a week, last dose taken within 24 hours prior to enrollment.

Inclusion Criteria for "CPAP-treated" Cohort:

* Diagnosis of OSA (based on home or attended sleep study) with an REI/AHI ≥ 15 with or without symptoms or REI/AHI ≥ 5 with symptoms of sleep apnea in a patient 18-85 years old.
* CPAP has been started within the last 2 years
* Patient is taking aspirin at a dose of 81mg/day for at least a week, last dose taken within 24 hours prior to enrollment.

Exclusion Criteria for all cohorts including control group:

* Patient is not able to provide informed consent
* Patient has taken at least one dose of a non-aspirin NSAID within the last 3 days
* Patient has taken at least one dose of another (non-aspirin) anti-platelet agent(s) (clopidogrel, abciximab, eptifibatide, tirofiban, cilostazol, dipyridamole, prasugrel, ticlopidine, ticagrelor) in the last 7 days.
* Patient has taken at least one dose of vitamin K antagonist (warfarin) in the last 7 days or heparin (low molecular weight or unfractionated) in the last 24 hours
* Patient has taken steroids (intravenous, oral, or topical) within the last 2 weeks
* Signs and symptoms of an active infection:
* Temperature ≥ 100.4
* Productive cough
* Rhinorrhea
* Dysuria
* Diarrhea
* Signs and symptoms of a local inflammatory reaction
* Pain
* Warmth
* Erythema
* Swelling
* Any history of a systemic inflammatory disorder
* Any history of diabetes mellitus if no HbA1C measurement obtained within 6 months is available; if HbA1C measurement obtained within 6 months is available, patient will be included.
* Any history of chronic kidney disease
* Pregnant women, and women in labor

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who come to the WCHN Pulmonary and Sleep Medicine Clinic either for a follow-up appointment to monitor their therapy for OSA or for an appointment to discuss a new diagnosis of OSA referred by their pulmonologist.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
The prevalence of aspirin resistance in patients with newly diagnosed OSA taking aspirin for primary or secondary prevention. | Immediately after consent is obtained (baseline)
  The prevalence of aspirin resistance, measured by platelet aggregometry, in patients with newly diagnosed OSA who take aspirin for primary or secondary prevention.

SECONDARY OUTCOMES:
The prevalence of aspirin resistance in OSA patients who take aspirin for primary or secondary prevention and are currently being treated with CPAP. | Immediately after consent is obtained (baseline)
  The prevalence of aspirin resistance in those patients with OSA on aspirin for primary or secondary prevention who are currently being treated with CPAP.

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Mendez, Principal Investigator — Nuvance Health
Locations (1):
- Danbury Hospital, Danbury, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peppard PE, Young T, Barnet JH, Palta M, Hagen EW, Hla KM. Increased prevalence of sleep-disordered breathing in adults. Am J Epidemiol. 2013 May 1;177(9):1006-14. doi: 10.1093/aje/kws342. Epub 2013 Apr 14. PMID 23589584
- [Background] Jordan AS, McSharry DG, Malhotra A. Adult obstructive sleep apnoea. Lancet. 2014 Feb 22;383(9918):736-47. doi: 10.1016/S0140-6736(13)60734-5. Epub 2013 Aug 2. PMID 23910433
- [Background] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Background] Maeder MT, Schoch OD, Rickli H. A clinical approach to obstructive sleep apnea as a risk factor for cardiovascular disease. Vasc Health Risk Manag. 2016 Mar 21;12:85-103. doi: 10.2147/VHRM.S74703. eCollection 2016. PMID 27051291
- [Background] Tazbirek M, Slowinska L, Kawalski M, Pierzchala W. The rheological properties of blood and the risk of cardiovascular disease in patients with obstructive sleep apnea syndrome (OSAS). Folia Histochem Cytobiol. 2011;49(2):206-10. doi: 10.5603/fhc.2011.0028. PMID 21744318
- [Background] Oga T, Chin K, Tabuchi A, Kawato M, Morimoto T, Takahashi K, Handa T, Takahashi K, Taniguchi R, Kondo H, Mishima M, Kita T, Horiuchi H. Effects of obstructive sleep apnea with intermittent hypoxia on platelet aggregability. J Atheroscler Thromb. 2009;16(6):862-9. doi: 10.5551/jat.2188. Epub 2009 Dec 22. PMID 20032579
- [Background] Kuliczkowski W, Witkowski A, Polonski L, Watala C, Filipiak K, Budaj A, Golanski J, Sitkiewicz D, Pregowski J, Gorski J, Zembala M, Opolski G, Huber K, Arnesen H, Kristensen SD, De Caterina R. Interindividual variability in the response to oral antiplatelet drugs: a position paper of the Working Group on antiplatelet drugs resistance appointed by the Section of Cardiovascular Interventions of the Polish Cardiac Society, endorsed by the Working Group on Thrombosis of the European Society of Cardiology. Eur Heart J. 2009 Feb;30(4):426-35. doi: 10.1093/eurheartj/ehn562. Epub 2009 Jan 27. PMID 19174428
- [Background] Cai G, Zhou W, Lu Y, Chen P, Lu Z, Fu Y. Aspirin resistance and other aspirin-related concerns. Neurol Sci. 2016 Feb;37(2):181-9. doi: 10.1007/s10072-015-2412-x. Epub 2015 Nov 14. PMID 26573589
- [Background] Gum PA, Kottke-Marchant K, Welsh PA, White J, Topol EJ. A prospective, blinded determination of the natural history of aspirin resistance among stable patients with cardiovascular disease. J Am Coll Cardiol. 2003 Mar 19;41(6):961-5. doi: 10.1016/s0735-1097(02)03014-0. PMID 12651041
- [Background] Lee PY, Chen WH, Ng W, Cheng X, Kwok JY, Tse HF, Lau CP. Low-dose aspirin increases aspirin resistance in patients with coronary artery disease. Am J Med. 2005 Jul;118(7):723-7. doi: 10.1016/j.amjmed.2005.03.041. PMID 15989905
- [Background] Grinstein J, Cannon CP. Aspirin resistance: current status and role of tailored therapy. Clin Cardiol. 2012 Nov;35(11):673-81. doi: 10.1002/clc.22031. Epub 2012 Jun 27. PMID 22740110
- [Background] Cheng G, Shan J, Xu G, Liu P, Zhou Y, Zhu Y, Lu X. Relationship between endothelial dysfunction, oxidant stress and aspirin resistance in patients with stable coronary heart disease. J Clin Pharm Ther. 2007 Jun;32(3):287-92. doi: 10.1111/j.1365-2710.2007.00823.x. PMID 17489881
- [Background] Hopps E, Caimi G. Obstructive Sleep Apnea Syndrome: Links Betwen Pathophysiology and Cardiovascular Complications. Clin Invest Med. 2015 Dec 4;38(6):E362-70. doi: 10.25011/cim.v38i6.26199. PMID 26654519
- [Background] Barbe F, Duran-Cantolla J, Sanchez-de-la-Torre M, Martinez-Alonso M, Carmona C, Barcelo A, Chiner E, Masa JF, Gonzalez M, Marin JM, Garcia-Rio F, Diaz de Atauri J, Teran J, Mayos M, de la Pena M, Monasterio C, del Campo F, Montserrat JM; Spanish Sleep And Breathing Network. Effect of continuous positive airway pressure on the incidence of hypertension and cardiovascular events in nonsleepy patients with obstructive sleep apnea: a randomized controlled trial. JAMA. 2012 May 23;307(20):2161-8. doi: 10.1001/jama.2012.4366. PMID 22618923
- [Background] Buchner NJ, Sanner BM, Borgel J, Rump LC. Continuous positive airway pressure treatment of mild to moderate obstructive sleep apnea reduces cardiovascular risk. Am J Respir Crit Care Med. 2007 Dec 15;176(12):1274-80. doi: 10.1164/rccm.200611-1588OC. Epub 2007 Aug 2. PMID 17673692
- [Background] Sokucu SN, Ozdemir C, Dalar L, Karasulu L, Aydin S, Altin S. Complete blood count alterations after six months of continuous positive airway pressure treatment in patients with severe obstructive sleep apnea. J Clin Sleep Med. 2014 Aug 15;10(8):873-8. doi: 10.5664/jcsm.3958. PMID 25126033
- [Background] Varol E, Ozturk O, Yucel H, Gonca T, Has M, Dogan A, Akkaya A. The effects of continuous positive airway pressure therapy on mean platelet volume in patients with obstructive sleep apnea. Platelets. 2011;22(7):552-6. doi: 10.3109/09537104.2011.578182. Epub 2011 May 19. PMID 21591980
- [Background] Krasopoulos G, Brister SJ, Beattie WS, Buchanan MR. Aspirin "resistance" and risk of cardiovascular morbidity: systematic review and meta-analysis. BMJ. 2008 Jan 26;336(7637):195-8. doi: 10.1136/bmj.39430.529549.BE. Epub 2008 Jan 17. PMID 18202034
- [Background] Schwammenthal Y, Tsabari R, Shenkman B, Schwartz R, Matetzky S, Lubetsky A, Orion D, Israeli-Korn S, Chapman J, Savion N, Varon D, Tanne D. Aspirin responsiveness in acute brain ischaemia: association with stroke severity and clinical outcome. Cerebrovasc Dis. 2008;25(4):355-61. doi: 10.1159/000118382. Epub 2008 Feb 28. PMID 18305387
- [Background] Ozben S, Ozben B, Tanrikulu AM, Ozer F, Ozben T. Aspirin resistance in patients with acute ischemic stroke. J Neurol. 2011 Nov;258(11):1979-86. doi: 10.1007/s00415-011-6052-7. Epub 2011 Apr 21. PMID 21509427
- [Background] Pasala T, Hoo JS, Lockhart MK, Waheed R, Sengodan P, Alexander J, Gandhi S. Aspirin Resistance Predicts Adverse Cardiovascular Events in Patients with Symptomatic Peripheral Artery Disease. Tex Heart Inst J. 2016 Dec 1;43(6):482-487. doi: 10.14503/THIJ-14-4986. eCollection 2016 Dec. PMID 28100965